CLINICAL TRIAL: NCT00076648
Title: A Phase III, Randomized, Controlled, Open-Label, Multicenter, Parallel Group Study Using Provisions for Exception From Informed Consent Requirements Designed to Evaluate the Safety and Efficacy of Poly SFH-P Injection [Polymerized Human Hemoglobin (Pyridoxylated), PolyHeme(R)] When Used to Treat Patients in Hemorrhagic Shock Following Traumatic Injuries Beginning in the Prehospital Setting
Brief Title: Safety and Efficacy of PolyHeme(R) in Hemorrhagic Shock Following Traumatic Injuries Beginning in the Pre-Hospital Setting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northfield Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTBSE-11-(N)
Record Dates: First submitted 2004-01-28; First posted 2004-01-30 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: Hemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — polyhemoglobin-pyridoxal-5-phosphate

INTERVENTIONS:
Drug: Poly SFH-P Injection

SUMMARY:
This study is designed to assess the survival benefit of administering PolyHeme to severely injured trauma patients in hemorrhagic shock beginning in the prehospital setting, where blood is not available, and continuing throughout a 12-hour postinjury hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients following trauma who have sustained blood loss and are in shock

Exclusion Criteria:

* Patients who have sustained unsurvivable injuries
* Patients who have severe head injury
* Pregnant females
* Patients found in cardiac arrest
* Patients who object to participation (e.g., religious grounds, wearing exclusion bracelet).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Scripps Mercy, San Diego, California
  - UC San Diego Medical Center, San Diego, California
  - Denver Health Medical Center, Denver, Colorado
  - Christiana Hospital, Newark, Delaware
  - Medical Center of Central Georgia, Macon, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - The Mayo Clinic, Rochester, Minnesota
  - Albany Medical Center, Albany, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Regional Resource Trauma Center, Bethlehem, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Johnson City Medical Center, Johnson City, Tennessee
  - University of Tennessee-Memphis, Memphis, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Memorial-Hermann Hospital, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - West Virginia University/Jon Michael Moore Trauma Center, Morgantown, West Virginia

REFERENCES:
- [Derived] Moore EE, Moore FA, Fabian TC, Bernard AC, Fulda GJ, Hoyt DB, Duane TM, Weireter LJ Jr, Gomez GA, Cipolle MD, Rodman GH Jr, Malangoni MA, Hides GA, Omert LA, Gould SA; PolyHeme Study Group. Human polymerized hemoglobin for the treatment of hemorrhagic shock when blood is unavailable: the USA multicenter trial. J Am Coll Surg. 2009 Jan;208(1):1-13. doi: 10.1016/j.jamcollsurg.2008.09.023. Epub 2008 Nov 7. PMID 19228496